CLINICAL TRIAL: NCT03356925
Title: Feasibility, Accuracy, and Effect of Point-of-care Xpert MTB/RIF Ultra and Xpert MTB/RIF Ultra Testing in Patients Suspected of Having TB: a Randomised Controlled Trial
Brief Title: Improving TB Diagnosis and Treatment Through Basic, Applied and Health Systems Research
Acronym: BAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Grant Theron, Associate Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N14/10/13
Record Dates: First submitted 2017-10-26; First posted 2017-11-29 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Tuberculosis
Keywords: Xpert®MTB/RIF; Xpert®MTB/RIF Ultra
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centralised Xpert®Ultra testing (No Intervention): Patients are selected to receive the standard of care for TB diagnosis at a centralised laboratory facility
- Xpert Ultra Point of Care testing (Active Comparator): Patients are selected to receive the point of care for TB diagnosis at the clinic facility they are visiting
  Interventions: Diagnostic Test: Xpert Ultra Point of Care testing

INTERVENTIONS:
Diagnostic Test: Xpert Ultra Point of Care testing — The intervention is the point of care Xpert Ultra TB diagnostic compared to the standard of care centralised TB testing at a centralised facility
  Arms: Xpert Ultra Point of Care testing

SUMMARY:
TB is a global health problem and in South Africa rates as the second most important problem in terms of Burden of Disease. There are many reasons for this, among which are diagnostic difficulties, extended treatments, drug resistance and health care provision. This application is concerned with all these drivers and will focus activities on a clinic which provides basic care in a very deprived socio-economic area of greater Cape Town, South Africa.

Patients studied in routine, but demanding environments are our focus as these clinics are representative of many areas where TB (and HIV) are found at high prevalence. If the constraints of working in such areas can be understood and appropriate changes that work made, the investigators believe the outputs and policy changes generated in this study will contribute to future success in other settings.

The investigators wish to study the implementation of the Xpert®MTB/RIF (Xpert) and Xpert Ultra (Ultra) systems in situ using a randomised controlled trial design, as opposed to a remote site (central laboratory), to assess whether time to diagnosis can be improved using point of care (POC). The investigators wish to maximise this opportunity by collecting biological samples from a patient population experiencing a TB epidemic for the evaluation of future TB diagnostics.

Using human DNA, the investigators will attempt to determine reasons for poor or no treatment response. Two possibilities exist for this: a) the M. tuberculosis strain is resistant to the drug in question or b) the patient is highly susceptible to the bacterium. The investigators will determine the exome sequences of study participants with susceptible M. tuberculosis strains who show poor or no response, and compare this with rapid responders. Using 16S rRNA sequencing, the investigators will also observe how the microbiome of TB patients is altered during TB treatment and how this is associated with treatment outcome, as well as after TB treatment.

This project will set the foundation for the implementation of new POC TB diagnostic technologies in clinics in South Africa. The biobanked specimens collected can be rapidly utilised for nascent technologies. Studying the patient microbiome will provide insights into what makes some patients more susceptible to TB and what microbiological changes occur during the course of anti-TB treatment.

DETAILED DESCRIPTION:
In 2015, the World Health Organization (WHO) estimated that there were there were an estimated 10.4 million new TB cases, 1.8 million deaths, and 580 000 cases of drug-resistant TB with 1.4 million deaths from TB among human immunodeficiency virus (HIV) negative people, and an additional 0.40 million deaths from HIV-associated TB. The African Region has approximately one quarter of the world's cases, and the highest rates of cases and deaths relative to population. The proportion of TB cases co-infected with HIV was highest in countries in the African Region; overall, 33% of TB cases were estimated to be co-infected with HIV in this region. South Africa is one of the countries with the highest number of incident cases in 2011 (410,000 - 600,000) making it one of the 22 high burden countries. Current estimates suggest that 330,000 of the incident cases are co-infected with HIV. Despite being declared an emergency in 1996 and the implementation of Direct Observed Therapy Short courses (DOTS) the case detection rate remains below the WHO target of 85%.

The DOTS strategy is promoted by the WHO as the optimal program to control the TB epidemic. According to the WHO, antibiotic treatment is effective in about 90% of patient, however, the duration of treatment places an enormous burden on health care services and patients often stop taking the treatment once the symptoms have improved. This implies that it is extremely challenging for TB control programmes to reach the WHO's target of 85% successful treatment. It is hypothesized that shortening the duration of treatment will significantly impact on adherence as well as treatment outcome. However therapeutic options are extremely limited given that there has been little antibiotic development over the past 40 years. The situation with respect to antibiotic resistant TB is considerably worse. Recent molecular epidemiological studies have provided convincing evidence that MDR-TB in South Africa is caused mostly by the transmission of MDR strains, as demonstrated by well-documented clonal outbreaks and elevated rates of primary resistance (in some places as high as 80%) among MDR-TB cases.

One of the effective means of combating drug resistant TB is the rapid diagnosis of any person with TB and detection of any potentially drug resistant TB strains in the early stages of the disease. Smear microscopy remains the state of the art diagnostic in many developing countries, but this method shows poor sensitivity which is further compromised by HIV co-infection. Culture-based methods remain the gold standard but are time consuming often leading to extensive diagnostic delays.

The WHO has called for expanding access to M. tuberculosis culture and drug susceptibility testing (DST) as part of the WHO Global laboratory strategic plan. Accordingly, 50% of the global population should have gained access to culture and DST services by 2010 and the scale-up should be completed by 2015, covering more than 5 billion people. But even if the access to culture and culture-based DST can be expanded in resource-poor settings, the slow turn-around time (several weeks) of culture-based DST limits the impact it has on treatment decisions and patient outcomes. This is especially true for HIV-infected TB suspects and children in whom a treatment decision should not be delayed due to rapid progression of disease and high risk of early mortality.

In June 2008, the WHO recommended the use of line probe assay (LPA) for rapid detection of MDR-TB in smear positive sputum specimens. These LPAs use polymerase chain reaction (PCR) to amplify regions of interest in the mycobacterial genome followed by reverse hybridization to sequence specific probes. The most prominent commercial DST product is the GenoType® MTBDRplus assay (HAIN Lifescience, GmbH, Nehren, Germany) for use in smear positive sputum samples or culture isolates. Both methods detect M. tuberculosis complex infection as well as mutations which cause RIF resistance (rpoB gene). The MTBDRplus assay can detect INH resistance by analysing the katG gene and the inhA promoter gene region. The sensitivity and specificity to detect INH and RIF resistance using the Genotype MTBDRplus has been shown to be high. In 2013, the Genotype MTBDRsl was endorsed by the WHO. This second line LPA assay allows the detection of resistance to fluoroquinolones, aminoglycosides, CAP, and EMB by targeting the gyrA, rrs and embB genes in M. tuberculosis, respectively. The sensitivity of the Genotype MTBDRsl ranges from 75 to 91% for detection of fluoroquinolone resistance, 77 to 85% for KANA resistance, 80 to 87% for CAP resistance, and 57 to 69% for EMB resistance.

There are some limitations to this technology. Firstly, not all the genotypes conferring resistance are known and secondly, DST methods are not all standardized and vary in their performance. This may result in suboptimal and variable sensitivities of the molecular based methods for certain drugs. The open-tube format of the method also allows for potential amplicon cross-contamination, which may lead to incorrect diagnoses and subsequent mismanagement of patients. Thus expensive infrastructure is required to enable these tests to be run.

An alternative diagnostics and DST solution became available in December 2010, when the WHO recommended the use of Xpert®MTB/RIF (Xpert), a closed, fully integrated and automated nested real-time PCR assay for rapid and simultaneous detection of M. tuberculosis complex and RIF resistance, for use as the first diagnostic test in TB suspects at risk of MDR-TB and HIV-associated TB. The method allows sample decontamination, PCR and real-time analysis to occur within a single disposable plastic cartridge. The turnaround time is less than 2 hours. The Xpert performs well for smear positive specimens, and shows promise for improving the diagnosis of smear-negative and extrapulmonary TB and RIF resistant TB specimens. Thus, this system may prove especially useful in settings where co-infection rates with HIV are high. However, the Xpert assay only has a ~70% sensitivity for detecting TB in smear negative samples and only provides information on RIF resistance. Furthermore, if the test indicates RIF resistance the specimen needs to be sent for second-line DST. Thus, the time gained by the rapid test is lost by the need for conventional DST tests. In addition, the test does not provide pharmacogenetic information which may be essential for formulation of an appropriate treatment regimen. Recently, the WHO has endorsed Xpert Ultra (Ultra), the successor of Xpert®MTB/RIF. Ultra retains its ability to detect rifampicin resisitance and is reported to be ten times more sensitive than its Xpert®MTB/RIF predecessor with total run-time for the nearly halved.

Xpert and MDRplus have been successfully implemented in the South African National Health Laboratory Service (NHLS). The NHLS implemented MTBDRplus LPA in 2008 with the aim to reduce the time to the initiation of treatment as compared to culture-based diagnostics. Despite a laboratory turnaround time of <7 days, the time to initiation of treatment was on average 55 days when MDR-TB was diagnosed. Examination of the cause of the additional delay showed that the laboratory turnaround time was significantly reduced but remained at 22 days for smear positive samples and 29 days for smear negative samples. This was explained by the high volume of samples needing testing and subsequent evaluation of the tests before distribution to the clinics. This highlights the need for re-tooling of the diagnostic laboratory to rapidly process and disseminate genetic-based tests. In addition, this study also highlighted the need to improve health systems to respond to rapid genetic based tests. No change was observed in the time between sending the diagnostic report and initiation of treatment (average 21 days, irrespective of the diagnostic method.

It is known that diagnostics in TB is difficult, but central to the control programme. Despite recent advances, diagnostics are not yet sufficiently rapid, cheap and comprehensive and even the introduction of the Xpert instrument has not dramatically reduced time to diagnosis or presumably patient retention. In South Africa, Xpert was introduced and scaled up rapidly in an attempt to address the TB epidemic, however, the testing equipment is centrally located.

The investigators propose a study which implements Xpert®MTB/RIF and Xpert Ultra for the testing of TB in symptomatic patients at the POC which could potentially improve the time-to-diagnosis and thus improve time to treatment initiation compared to centralised testing.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing to provide specimens (urine, blood, stool, respiratory tract specimens and swabs)
* The patient is clinically suspected of having TB (Two WHO TB symptoms for HIV negative patients and one WHO TB symptom if HIV positive)

Exclusion Criteria:

* The patient is under the age of 18 years old
* The patient declines consent
* The patient has too few clinical symptoms for TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1549 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Treatment time | Up to 8 weeks
  Time-specific proportion of patients starting TB treatment (all patients and confirmed cases) in centralised diagnosis and treatment arm compared to POC arm.

SECONDARY OUTCOMES:
TB diagnosis time | Up to 8 weeks
  Time-specific proportion of patients diagnosed in centralised vs POC arm
Time specific yield of Xpert Ultra | Up to 8 weeks
  Proportion of patients who are Xpert Ultra positive
Airway and gut microbiome composition before, during, and after TB treatment | Up to 18 months
  Microbial composition determined by next-generation sequencing of bacterial DNA in respiratory tract specimens and stool

CONTACTS AND LOCATIONS:
Overall Officials: Grant Theron, PhD, Principal Investigator — University of Stellenbosch
Locations (2):
- South Africa (2):
  - Scottsdene Clinic, Cape Town, Western Cape
  - Wallacedene Clinic, Cape Town, Western Cape

REFERENCES:
- [Background] Theron G, Zijenah L, Chanda D, Clowes P, Rachow A, Lesosky M, Bara W, Mungofa S, Pai M, Hoelscher M, Dowdy D, Pym A, Mwaba P, Mason P, Peter J, Dheda K; TB-NEAT team. Feasibility, accuracy, and clinical effect of point-of-care Xpert MTB/RIF testing for tuberculosis in primary-care settings in Africa: a multicentre, randomised, controlled trial. Lancet. 2014 Feb 1;383(9915):424-35. doi: 10.1016/S0140-6736(13)62073-5. Epub 2013 Oct 28. PMID 24176144
- [Background] Johnson R, Warren R, Strauss OJ, Jordaan AM, Falmer AA, Beyers N, Schaaf HS, Murray M, Cloete K, van Helden PD, Victor TC. An outbreak of drug-resistant tuberculosis caused by a Beijing strain in the western Cape, South Africa. Int J Tuberc Lung Dis. 2006 Dec;10(12):1412-4. PMID 17167961
- [Background] Petti CA, Polage CR, Quinn TC, Ronald AR, Sande MA. Laboratory medicine in Africa: a barrier to effective health care. Clin Infect Dis. 2006 Feb 1;42(3):377-82. doi: 10.1086/499363. Epub 2005 Dec 20. PMID 16392084
- [Background] Detjen AK, DiNardo AR, Leyden J, Steingart KR, Menzies D, Schiller I, Dendukuri N, Mandalakas AM. Xpert MTB/RIF assay for the diagnosis of pulmonary tuberculosis in children: a systematic review and meta-analysis. Lancet Respir Med. 2015 Jun;3(6):451-61. doi: 10.1016/S2213-2600(15)00095-8. Epub 2015 Mar 24. PMID 25812968
- [Background] Theron G, Peter J, Dowdy D, Langley I, Squire SB, Dheda K. Do high rates of empirical treatment undermine the potential effect of new diagnostic tests for tuberculosis in high-burden settings? Lancet Infect Dis. 2014 Jun;14(6):527-32. doi: 10.1016/S1473-3099(13)70360-8. Epub 2014 Jan 15. PMID 24438820
- [Background] Marais BJ, Brittle W, Painczyk K, Hesseling AC, Beyers N, Wasserman E, van Soolingen D, Warren RM. Use of light-emitting diode fluorescence microscopy to detect acid-fast bacilli in sputum. Clin Infect Dis. 2008 Jul 15;47(2):203-7. doi: 10.1086/589248. PMID 18532893
- [Background] Ling DI, Zwerling AA, Pai M. GenoType MTBDR assays for the diagnosis of multidrug-resistant tuberculosis: a meta-analysis. Eur Respir J. 2008 Nov;32(5):1165-74. doi: 10.1183/09031936.00061808. Epub 2008 Jul 9. PMID 18614561
- [Background] Hillemann D, Rusch-Gerdes S, Richter E. Feasibility of the GenoType MTBDRsl assay for fluoroquinolone, amikacin-capreomycin, and ethambutol resistance testing of Mycobacterium tuberculosis strains and clinical specimens. J Clin Microbiol. 2009 Jun;47(6):1767-72. doi: 10.1128/JCM.00081-09. Epub 2009 Apr 22. PMID 19386845
- [Background] Kiet VS, Lan NT, An DD, Dung NH, Hoa DV, van Vinh Chau N, Chinh NT, Farrar J, Caws M. Evaluation of the MTBDRsl test for detection of second-line-drug resistance in Mycobacterium tuberculosis. J Clin Microbiol. 2010 Aug;48(8):2934-9. doi: 10.1128/JCM.00201-10. Epub 2010 Jun 23. PMID 20573868
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Boehme CC, Nicol MP, Nabeta P, Michael JS, Gotuzzo E, Tahirli R, Gler MT, Blakemore R, Worodria W, Gray C, Huang L, Caceres T, Mehdiyev R, Raymond L, Whitelaw A, Sagadevan K, Alexander H, Albert H, Cobelens F, Cox H, Alland D, Perkins MD. Feasibility, diagnostic accuracy, and effectiveness of decentralised use of the Xpert MTB/RIF test for diagnosis of tuberculosis and multidrug resistance: a multicentre implementation study. Lancet. 2011 Apr 30;377(9776):1495-505. doi: 10.1016/S0140-6736(11)60438-8. Epub 2011 Apr 18. PMID 21507477
- [Background] Theron G, Peter J, van Zyl-Smit R, Mishra H, Streicher E, Murray S, Dawson R, Whitelaw A, Hoelscher M, Sharma S, Pai M, Warren R, Dheda K. Evaluation of the Xpert MTB/RIF assay for the diagnosis of pulmonary tuberculosis in a high HIV prevalence setting. Am J Respir Crit Care Med. 2011 Jul 1;184(1):132-40. doi: 10.1164/rccm.201101-0056OC. Epub 2011 Apr 14. PMID 21493734
- [Background] Warren RM, Streicher EM, Gey van Pittius NC, Marais BJ, van der Spuy GD, Victor TC, Sirgel F, Donald PR, van Helden PD. The clinical relevance of Mycobacterial pharmacogenetics. Tuberculosis (Edinb). 2009 May;89(3):199-202. doi: 10.1016/j.tube.2009.03.001. Epub 2009 May 1. PMID 19409848
- [Background] Jacobson KR, Theron D, Kendall EA, Franke MF, Barnard M, van Helden PD, Victor TC, Streicher EM, Murray MB, Warren RM. Implementation of genotype MTBDRplus reduces time to multidrug-resistant tuberculosis therapy initiation in South Africa. Clin Infect Dis. 2013 Feb;56(4):503-8. doi: 10.1093/cid/cis920. Epub 2012 Oct 22. PMID 23090928
- [Background] Theron G, Peter J, Calligaro G, Meldau R, Hanrahan C, Khalfey H, Matinyenya B, Muchinga T, Smith L, Pandie S, Lenders L, Patel V, Mayosi BM, Dheda K. Determinants of PCR performance (Xpert MTB/RIF), including bacterial load and inhibition, for TB diagnosis using specimens from different body compartments. Sci Rep. 2014 Jul 11;4:5658. doi: 10.1038/srep05658. PMID 25014250
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229
- See also: WHO Global tuberculosis report 2016 — http://apps.who.int/iris/bitstream/10665/250441/1/9789241565394-eng.pdf
- See also: WHO Global tuberculosis report 2012 — http://apps.who.int/iris/bitstream/10665/75938/1/9789241564502_eng.pdf
- See also: WHO Xpert MTB/RIF implementation manual 2014 — http://apps.who.int/iris/bitstream/10665/112469/1/9789241506700_eng.pdf
- See also: WHO Expert group meeting report. The use of molecular line probe assay for the detection of resistance to second-line anti-tuberculosis drugs. 2013 — http://apps.who.int/iris/bitstream/10665/78099/1/WHO_HTM_TB_2013.01.eng.pdf